CLINICAL TRIAL: NCT00569140
Title: A Phase 1, Single Ascending Dose Trial to Establish the Safety, Tolerability and Pharmacokinetic Profile of Intravitreous Injections of E10030 (Anti-PDGF Pegylated Aptamer) Monotherapy and of E10030 Given in Combination With Lucentis®0.5 Mg/Eye in Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: A Phase 1, Safety, Tolerability and Pharmacokinetic Profile of Intravitreous Injections of E10030 (Anti-PDGF Pegylated Aptamer) in Subjects With Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Denise Teuber, Ophthotech Corp
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPH 1000
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2010-01

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — E10030 aptamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention): E10030
  Interventions: Drug: E10030

INTERVENTIONS:
Drug: E10030 — Intravitreal injection

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability, and pharmacokinetic profile of E10030 intravitreous injection when administered as monotherapy or in combination with Lucentis® 0.5 mg/eye in subjects with subfoveal choroidal neovascularization secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

Subfoveal choroidal neovascularization (CNV) due to AMD

Exclusion Criteria:

* Any of the following underlying diseases including:

  * Diabetic retinopathy.
  * History or evidence of severe cardiac disease (e.g., NYHA Functional Class III or IV - see Appendix 19.6), history or clinical evidence of unstable angina, acute coronary syndrome, myocardial infarction or revascularization with 6 months, ventricular tachyarrythmias requiring ongoing treatment.
  * History or evidence of clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation.
  * Clinically significant impaired renal (serum creatinine >2.5 mg/dl or s/p renal transplant or receiving dialysis) or hepatic function.
  * Stroke (within 12 months of trial entry).
  * Any major surgical procedure within one month of trial entry. Previous therapeutic radiation in the region of the study eye. Any treatment with an investigational agent in the past 60 days for any condition.

Known serious allergies to the fluorescein dye used in angiography, to the components of the ranibizumab formulation, or to the components of the E10030 formulation.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-12; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Ophthalmic DLTs | immediate

SECONDARY OUTCOMES:
adverse events | immendiate

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Teuber, New York, New York, United States